CLINICAL TRIAL: NCT07292285
Title: The Surveillance Nonoperative Watch & Wait (SNOWW) Rectal Cancer Trial
Acronym: SNOWW
Status: Not yet recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 25-1647.cc
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cancer of the Rectum
Keywords: Management of Stage 2 or 3 Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ctDNA testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rectal Cancer Clinical Stage II or III

SUMMARY:
The primary objectives of this study are to determine if the inclusion of ctDNA testing in the evaluation and management of stages 2 and 3 rectal cancers will allow clinicians to improve their selection of patients for wait and watch (WW) management and to facilitate the detection of cancer regrowth during WW surveillance.

DETAILED DESCRIPTION:
This will be a prospective multi-center observational study for adult patients with stage 2 or 3 rectal adenocarcinoma who will be treated with TNT and are potential candidates for WW management. Study eligibility will be determined prior to the initiation of TNT by individual site investigators with the expectation that both the patient and investigator will be involved in multidisciplinary cancer decision-making. The rectal cancer tissue samples that were used to make the cancer diagnosis will also be used by our collaborative sponsor (Natera, Inc) to develop a tissue-informed and patient-specific ctDNA profile for each study patient. Patient blood samples will then be collected before the start of TNT, during TNT, after the completion of TNT, and for WW patients, at the time of every scheduled endoscopic surveillance exam, as recommended by the NCCN, and when non-scheduled endoscopic exams are performed. Figure 1. The patients will be prospectively followed for 2 years after the initiation of W&W or until cancer regrowth is suspected or confirmed and treatments other than WW are implemented. Patients who have cancer regrowth and then salvage surgery will be followed until their first postoperative cancer re-staging examination. Patients who have cancer regrowth and do not have salvage surgery will be followed. until this decision to not pursue salvage surgery is made.

The study surgeons and their patients will have access to their ctDNA test results. The study surgeon and other members of the patients' cancer care team will be advised to consider these results in their patient care decision-making and to document how each ctDNA effected decision making, if at all. The study surgeon will be responsible for ensuring that their patients are aware of the limitations of ctDNA testing and the NCCN recommendations for its use in WW management of rectal cancer.

To evaluate the impact of ctDNA on the shared decision-making process, the validated 9 Item Shared Decision-Making Questionnaire (SDM-Q-9) and the Control Preference Sale (CPS) will be administered to patients at the re-staging visit following TNT, when the decision to pursue WW or surgery is being considered. For patients managed with WW, the SDM-Q-9 will also be re-administered every time ctDNA is used in surveillance and whether a treatment decision is being actively reconsidered based on ctDNA results.

Additionally, the Shared Decision-Making Questionnaire- Physician Version (SDM-Q-Doc) will be completed by study surgeons at the re-staging visit following TNT, when the decision to pursue WW or surgery is being considered. For patients managed with WW, the SDM-Q-Doc will also be re-administered every time ctDNA is used in surveillance and whether a treatment decision is being actively reconsidered based on ctDNA results. This will allow assessment of surgeon perspectives on the decision-making process and how ctDNA influences clinical recommendations

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.

Additional Inclusion Criteria:

Pre-TNT phase Adult male and female patients (>18 years old) Clinical stage 2 or 3 rectal cancer, within or beyond the reach of digital rectal exam (DRE), who are evaluated in a multidisciplinary setting and who will receive induction or consolidation total neoadjuvant therapy (TNT) and are candidates for watch and wait management (WW) with curative intent.

Post-TNT phase complete or near complete clinical response to TNT High-definition flexible endoscopy: Pale smooth scar with or without telangiectasia No ulceration, nodularity, or mucosal irregularities No stricture DRE: Smooth, flat scar No nodularity Diffusion-weighted MRI2 Fibrotic, linear scar with low signal intensity on T2-weighted images No diffusion restriction No suspicious lymph nodes

Near Complete Clinical Response:

Endoscopic appearance with irregular small mucosal nodules, superficial ulceration, or mild persistent erythema DRE: Smooth induration or superficial minor mucosal irregularity MRI: T2-weighted MRI with downstaging with or without residual fibrosis, small area of residual signal, and complete or partial regression of lymph nodes. Diffusion-weighted MRI with small area of residual high signal intensity

Exclusion Criteria:

* • Patients who are less than 18 years old

  * Patients who are pregnant during the study period
  * Patients with stage I or IV rectal cancer
  * Patients who receive neoadjuvant therapy other than TNT.
  * Patients who receive short-course neoadjuvant radiotherapy.
  * Patients who are actively enrolled in other clinical trials that prohibit inclusion in this study.
  * Patients who refuse or are unable to undergo ctDNA testing and subsequent follow ups
  * Patients who refuse or are unable to undergo WW management of rectal cancer.
  * Patients who are undergoing "WW" management of rectal cancer due to refusal of recommended surgical resection. (For example, the hypothetical patient with an incomplete clinical response to TNT who refuses surgery).
  * Patients who undergo WW for palliation only.
  * Patients with prior history of rectal cancer with or without chemoradiation treatment or surgical resection
  * Patients who have a different cancer, in addition to rectal cancer, in whom the study ctDNA testing would be uninterpretable.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rectal Cancer Stage II or III
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Improve selection of patients for WW management | 36 months
  determine if the inclusion of ctDNA testing in the evaluation and management of stages 2 and 3 rectal cancers will allow clinicians to improve their selection of patients for WW management and to facilitate the detection of cancer regrowth during WW surveillance.

CONTACTS AND LOCATIONS:
Overall Officials: Jon MT Vogel, MD, Principal Investigator — University of Colorado Denver Anschutz Medical Campus

IPD SHARING:
Plan to Share IPD: No
A plan has not been put in place at this time